CLINICAL TRIAL: NCT06338163
Title: Polihexanide SSIs Measures Bundle (PSMB) During Enhanced Recovery After Major Digestive Surgery
Acronym: POSSIBLE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Marco Catarci (Other)
Collaborators: Associazione Chirurghi Ospedalieri Italiani (Other)
Responsible Party: Sponsor-Investigator, Marco Catarci, Study Chair, Ospedale Sandro Pertini, Roma
Organization: Ospedale Sandro Pertini, Roma (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POSSIBLE 1.6
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Surgical Site Infection; Surgical Procedures, Operative
Keywords: surgical site infection; polihexanide; preoperative decontamination
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Randomized controlled prospective multicenter
Who Masked: Outcomes Assessor
Masking Description: Assessor of the primary outcome will be masked concerning arm allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Once a day starting 5 days before the operation:
  Total body washing with usual soap/shampoo and single-use washcloths impregnated with a mix of Polihexanide, surfactants, and excipients.
  Nasal cleaning 3 times a day with a Polihexanide Nasal Gel Oral gargles 3 times a day using 10 mL of a Polihexanide oral solution. After the closure of fascia, 10 minutes subcutaneous irrigation with 50 to 250 mL (according to incision length) of antiseptic solution will be performed using a 0.04% sterile Polihexanide solution. After the end of the application time, a subcutaneous swab for culture will be taken. Before standard (according to local center clinical practice) wound(s) dressing(s), a 3 mm-thick antiseptic gel (a combination comprised of 0.1 % Polihexanide and 0.1 % propyl betaine (surfactant) that is used for cleansing, moistening and decontamination of post-operative wounds) will be applied on any wound(s).
  Interventions: Combination Product: Polihexanide-based bundle
- Control (Active Comparator): Once a day starting 5 days before the operation:
  Total body washing with usual soap/shampoo. No oral and nasal MDRO-decolonization will be performed. After the closure of fascia, 10 minutes subcutaneous irrigation with 50 to 250 mL (according to incision length) NS will be performed. After the end of the application time, a subcutaneous swab for culture will be taken. Finally, standard wound(s) dressing(s) (according to local center clinical practice) will be applied.
  Interventions: Combination Product: Standard bundle

INTERVENTIONS:
Combination Product: Polihexanide-based bundle — Pre- and intra-operative decontamination will be accomplished in the treatment (experimental) arm with Polihexanide-based products
  Other Names: Prontoderm® Wipes (B. Braun Medical AG, Sempach, Switzerland); Prontoderm® Nasal Gel (B. Braun Medical AG, Sempach, Switzerland); ProntOral® (B. Braun Medical AG, Sempach, Switzerland); LavaSurge® (B. Braun Medical AG, Sempach, Switzerland)
  Arms: Treatment
Combination Product: Standard bundle — Pre- and intra-operative decontamination will be accomplished in the control arm with normal soap/shampoo and saline solution
  Arms: Control

SUMMARY:
This is a randomized controlled, prospective, multicenter superiority trial with two parallel treatment groups and single blinding (local investigators performing postoperative follow up will be blinded for group allocation), with prospective enrollment planned from July 2024 to June 2025 in 20 Italian surgical centers. All patients undergoing elective major gastro-intestinal (GI) tract surgery (upper GI, HPB, & lower GI) will be included in a prospective database after written informed consent. A total of 2,000 patients is expected based on a mean of 100 cases per center.

DETAILED DESCRIPTION:
Just after signing a written informed consent to participate, patients will randomly be assigned either to the experimental group (Polihexanide bundle) or to the control group. Block randomization (blocks of 10 patients per single participating center) will be performed using an unstratified computer generated randomization list. All operations will be performed according to local criteria of the participating center. Hair removal will be accomplished on the day of surgery with electronic clippers. Alcohol-based solutions of chlorhexidine for surgical site skin preparation will be used. A first dose of perioperative i.v. antibiotics will be administered 30 minutes before skin incision (choice of the antibiotic according to local criteria) in all patients. Additional intraoperative doses will be administered for procedures exceeding two half-lives of the antibiotic. At the end of the operation, the peritoneal cavity will be rinsed routinely with 0.9% sodium chloride solution (normal saline, NS) at body temperature. Before closure of fascia, instruments and gloves will be changed. The eventual placement of drain(s) in the peritoneal cavity and/or creation of an intestinal stoma will be recorded. No subcutaneous suture or drainage will be done. Skin will be closed with either staples, intracutaneous running suture or interrupted sutures.

Potential patient-specific and intraoperative risk factors will be recorded: sex, age, body mass index, nutritional status, frailty, indication to surgery (benign vs. malignant disease), perioperative administration of steroids, renal failure and dialysis, cardiovascular or respiratory disease, American Society of Anesthesiologist class, bowel preparation, type of approach, operative time, presence of peritoneal cavity drainage. During the postoperative period, patients will be examined by the attending surgeon daily. Fever (central temperature > 38 °C), pulse, abdominal signs, bowel movements, volume and aspect of drainage (if present) will be recorded daily. The local attending surgeon will make any decision for complementary exams and imaging according to his own criteria. The rate of any adverse event will be calculated and graded according to the Clavien-Dindo criteria [19] and to Japan Clinical Oncology Group Postoperative Complications (JCOG-PC) extended criteria [20], including all anastomotic leaks, wound infection (according to the definitions of the Centers for Disease Control and Prevention and wound culture), pneumonia (clinical symptoms, and physical and radiological examinations), central venous line infection (positive blood culture), urinary tract infection (positive urine culture with bacterial count). ERAS pathway items will be defined according to national [27] guidelines, measuring adherence upon explicit criteria. All data will be recorded for a minimum of 8 weeks (60 days) after surgery. PROM questionnaires will be administered to all enrolled patients four to one week before the planned operation, at discharge, and 6 to 8 weeks after the operation.

After anonymization, all data of each single case will be prospectively uploaded by local investigator(s) on a web-based database, protected by individual access credentials, and incorporated into a spreadsheet for data analysis. Any eventual discrepancy and/or mismatch will be checked, addressed and solved through strict cooperation between coordinating and local investigators.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to laparoscopic/robotic/open/converted major digestive surgery (upper and lower gastrointestinal resections).
* American Society of Anesthesiologists' (ASA) class I, II, III or IV
* Elective surgery
* Patients' written acceptance to be included in the study.

Exclusion Criteria:

* American Society of Anesthesiologists' (ASA) class V
* Urgent surgery
* Pregnancy
* Hyperthermic intraperitoneal chemotherapy for carcinomatosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infections rate | 60 days after surgery
  CDC definition
Incisional (superficial and deep) Surgical Site Infections rate | 60 days after surgery
  CDC definition
Infectious morbidity rates | 60 days after surgery
  SSI + urinary tract infection + pulmonary infection

SECONDARY OUTCOMES:
Anastomotic leakage rates | 60 days after surgery
  According to international consensus
Overall morbidity rates | 60 days after surgery
  Any adverse event
Major morbidity rates | 60 days after surgery
  Any adverse event grade > II according to Clavien-Dindo
Comprehensive complication index | 60 days after surgery
  According to Slankamenac et al 2013
Overall length of postoperative hospital stay | 60 days after surgery
  inclusive of any unplanned readmission
Readmission rates | 60 days after surgery
  any unplanned readmission after primary discharge

OTHER OUTCOMES:
Patient-reported outcome measures | preoperative, at discharge, 60 days after surgery
  MD Anderson Symptom Inventory for Gastrointestinal Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marco Catarci, MD, FACS, Study Chair — Associazione Chirurghi Ospedalieri Italiani; Massimo Sartelli, MD, Principal Investigator — Ospedale di Macerata
Locations (3):
- Italy (3):
  - OSpedale Santa Maria Annunziata, Florence, FI
  - Ospedale Civile di Macerata, Macerata, MC
  - Ospedale Sandro Pertini, Roma, RM

IPD SHARING:
Plan to Share IPD: Undecided
complete dataset after study completion will be availble upon request

REFERENCES:
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Katayama H, Kurokawa Y, Nakamura K, Ito H, Kanemitsu Y, Masuda N, Tsubosa Y, Satoh T, Yokomizo A, Fukuda H, Sasako M. Extended Clavien-Dindo classification of surgical complications: Japan Clinical Oncology Group postoperative complications criteria. Surg Today. 2016 Jun;46(6):668-85. doi: 10.1007/s00595-015-1236-x. Epub 2015 Aug 20. PMID 26289837
- [Background] Strobel RM, Leonhardt M, Krochmann A, Neumann K, Speichinger F, Hartmann L, Lee LD, Beyer K, Daum S, Kreis ME, Lauscher JC. Reduction of Postoperative Wound Infections by Antiseptica (RECIPE)?: A Randomized Controlled Trial. Ann Surg. 2020 Jul;272(1):55-64. doi: 10.1097/SLA.0000000000003645. PMID 31599810
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- [Background] Allegranzi B, Bischoff P, de Jonge S, Kubilay NZ, Zayed B, Gomes SM, Abbas M, Atema JJ, Gans S, van Rijen M, Boermeester MA, Egger M, Kluytmans J, Pittet D, Solomkin JS; WHO Guidelines Development Group. New WHO recommendations on preoperative measures for surgical site infection prevention: an evidence-based global perspective. Lancet Infect Dis. 2016 Dec;16(12):e276-e287. doi: 10.1016/S1473-3099(16)30398-X. Epub 2016 Nov 2. PMID 27816413
- [Background] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Background] Mueller TC, Loos M, Haller B, Mihaljevic AL, Nitsche U, Wilhelm D, Friess H, Kleeff J, Bader FG. Intra-operative wound irrigation to reduce surgical site infections after abdominal surgery: a systematic review and meta-analysis. Langenbecks Arch Surg. 2015 Feb;400(2):167-81. doi: 10.1007/s00423-015-1279-x. Epub 2015 Feb 14. PMID 25681239